CLINICAL TRIAL: NCT02095470
Title: Advanced Video Laryngoscope, a New Practical Intubation Device: Randomized Clinical Trial in 401 Patients
Brief Title: Video Laryngoscope, New Intubation Device
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Education Development Center, Inc. (Industry)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 93-4678; 93-4687 (Other: shiraz university o medical sciences)
Record Dates: First submitted 2014-03-15; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Elective Intubation
Keywords: Laryngoscopy; Equipment; Video Laryngoscope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- videolaryngoscope group (Experimental): video laryngoscopy was done for them
  Interventions: Device: video laryngoscope
- traditional laryngoscope (Placebo Comparator): comparison to active group with routine laryngoscope
  Interventions: Device: traditional laryngoscope

INTERVENTIONS:
Device: video laryngoscope — newly developed innovatory device
  Other Names: glidescope
  Arms: videolaryngoscope group
Device: traditional laryngoscope — traditional way for intubation
  Arms: traditional laryngoscope

SUMMARY:
new glidoscope was tested on 401 patients

DETAILED DESCRIPTION:
Four hundred and one patients who were scheduled for elective operation, were randomly assigned to be intubated by direct laryngoscopy using a Macintosh blade size 3rd (DL, n=196) or intubation using the video laryngoscope (VL, n=205). Prior to intubation all patients were given a similar regimen of induction of anesthesia. The patients were then intubated, using direct laryngoscopy or the VL, by a different anesthetist during which the larynx was inspected and given a laryngoscopy score. Time to intubate, failure rate, injuries, personnel pleasure and, aspiration rate were measured

ELIGIBILITY:
Inclusion Criteria:

* elective operation who filled the consent

Exclusion Criteria:

* poor intubation
* emergency cases
* hemodynamic derangement

Ages: 19 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
laryngoscopy grade | hospital stay (average 48 hours)
  grade of laryngoscopy
time to intubation | 60 minutes
  time to successful intubation in minutes
unsuccessful attempts | 60 minutes
  number of failure

SECONDARY OUTCOMES:
aspiration | hospital stay ( 48 hours)
  clinical aspiration or radiological

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz Universty of Mesical Sciences, Shiraz, Fars, Iran